CLINICAL TRIAL: NCT03143699
Title: The Effect of Immediate Feedback on Long-term Blood Pressure Measurement Skills: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1.712.520
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-05

CONDITIONS: Education, Medical; Blood Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate feedback (Experimental): Submitted to a training on blood pressure measurement skills and an immediate feedback after their encounter with an standardized patient - SP
  Interventions: Other: Immediate Feedback
- Students with no immediate feedback (No Intervention): Submitted to a training on blood pressure measurement skills, but without an immediate feedback after their encounter with an standardized patient - SP

INTERVENTIONS:
Other: Immediate Feedback — Students will be trained to measure blood pressure in the same way, with a brief 4-hour theoretical-practical intervention. After the training, students will measure the blood pressure of a standardized patient and observers will evaluate them using a checklist. After that, students from the intervention group will receive an immediate feedback based on the previous literature. Briefly, feedback will be based on what was directly observed and will be phrased in non-judgmental language, following the Pendleton model.
  Arms: Immediate feedback

SUMMARY:
The present study aims to investigate the effect of immediate feedback on long-term blood pressure measurement skills. This is a randomized controlled trial including first year students from a Brazilian medical school, which will be randomized in two groups: an intervention group (submitted to a training on blood pressure measurement skills and an immediate feedback) and a control group (submitted to a training on blood pressure measurement skills, but with no immediate feedback). Then, students will be assessed 3 months after the feedback in order to see whether there will be a difference between groups. Our hypothesis is that students submitted to immediate feedback would have better scores in the blood-pressure measurement skills after 3 months. A knowledge questionnaire as well as a standardized patient scenario will be used to assess students' knowledge and skills.

DETAILED DESCRIPTION:
There are several studies evaluating the role of feedback in medical education, showing promising outcomes. Although, immediate feedback is associated with better knowledge and skills in short-term, few studies have assessed whether immediate feedback could impact the maintenance of skills. The present study aims to investigate the effect of immediate feedback on long-term blood pressure measurement skills. This is a randomized controlled trial including first year students from a Brazilian medical school, which will be randomized in two groups: an intervention group (submitted to a training on blood pressure measurement skills and an immediate feedback after their encounter with an standardized patient - SP) and a control group (submitted to the same training on blood pressure measurement skills, but with no immediate feedback after the SP encounter).

Both groups will be trained to measure blood pressure in the same way, with a brief 4-hour theoretical-practical intervention. After the training, students will measure the blood pressure of a standardized patient and observers will evaluate them using a checklist.

Then, students will have no other exposure to the BP training for three months and they will be invited again to participate in another SP encounter. Differences on BP skills after 3 months between those exposed to immediate feedback and those not exposed to immediate feedback would be investigated.

ELIGIBILITY:
Inclusion criteria:

* students officially registered in the first semester of the medical school and older than 18 years old.

Exclusion criteria:

* those absent in any part of the blood pressure measurement training and those who not signed the consent term

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-11-06 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Assess blood-pressure measurement skills | 3 months
  Blood pressure measurement skills checklist - following the criteria adopted by international (Eighth Joint National Committee) and the Brazilian guidelines (VII Brazilian Guidelines on Hipertension)

SECONDARY OUTCOMES:
Assess blood-pressure measurement knowledge | 3 months
  Blood pressure measurement knowledge test - following the criteria adopted by international (Eighth Joint National Committee) and the Brazilian guidelines (VII Brazilian Guidelines on Hipertension)

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Lucchetti, MD, PhD, Study Director — Federal University of Juiz de Fora
Locations (1):
- Faculdade de Ciências Médicas e da Saúde de Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No